CLINICAL TRIAL: NCT05990894
Title: Efficacy and Safety of Steroid for Treatment of Acute/Subacute Severe Cerebral Venous Thrombosis.
Brief Title: Steroid for Treatment of Acute/Subacute Severe Cerebral Venous Thrombosis.
Status: Completed | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, JiangangDuan, MD, PhD, Xuanwu Hospital, Beijing
Other Study IDs: [2020]098
Record Dates: First submitted 2023-08-06; First posted 2023-08-14 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Cerebral Venous Thrombosis
Keywords: Cerebral venous thrombosis; Severe cerebral venous thrombosis; Steroid therapy
MeSH Terms: conditions — Intracranial Thrombosis | interventions — Methylprednisolone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Standard treatment group: Each patient received subcutaneous low-molecular-weight heparin in adjusted doses for 10 to 14 days, followed by oral anticoagulants (warfarin or dabigatran or rivaroxaban, if warfarin was used, PT-INR was maintained between 2.0 and 3.0) for 6 months or more. The use of endovascular treatment (local thrombectomy/thrombolysis) was reserved for patients who are still progressing with adequate anticoagulant therapy.
- Steroid therapy group: Patients in the steroid therapy group received short-term steroids in addition to standard anticoagulant therapy.
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Methylprednisolone — In the steroid therapy group, patients received standard treatment plus steroid therapy. Steroid therapy protocol is as follows: 500 mg methylprednisolone once a day, intravenous drip for 3 days, then reduced to 80 mg once a day, intravenous drip for 5 days, and changed to oral methylprednisolone/prednisone 1 mg per kilogram body weight, gradually tapered off by a dose of 10 mg per week.
  Groups: Steroid therapy group

SUMMARY:
The cohort study aims to evaluate the efficacy and safety of steroids combined with anticoagulant therapy compared to standard anticoagulant therapy in acute/subacute severe cerebral venous thrombosis.

DETAILED DESCRIPTION:
Background: Evidence suggests that the inflammatory response plays a crucial role in regulating severe CVT pathogenesis. However, whether CVT patients can benefit from anti-inflammatory therapy has been debated.

Objective: The objective of this cohort study is to explore the efficacy and safety of steroids combined with anticoagulant therapy compared to standard anticoagulant therapy in acute/subacute severe cerebral venous thrombosis (CVT) patients.

Method: We reviewed the data of patients with acute/subacute severe CVT treated with a short-term application of steroid or not from a prospective stroke registry of our center. We compared functional outcomes and major adverse events at 6 months follow-up after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Acute or subacute severe CVT, determined by the onset-to-admission time (≤ 15 days) or symptom aggravation-to-admission time (≤ 15 days) and MRI+MRV/MRBTI (MR Black-Blood Thrombus Imaging), or CT+CTV

Exclusion Criteria:

* younger than 14 years；
* foreign nationality；
* receiving steroids before the onset of CVT；
* patients with other serious diseases；
* Presenting with neurological deficits before the onset of CVT；
* lack of baseline data before treatment；
* receiving steroids during hospitalization for other reasons but the dosage did not reach pulsed-therapy level
* brain herniation but refusing to undergo decompressive craniectomy, or pupillary light reflex did not recover after decompressive craniectomy

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients with acute/subacute severe CVT were enrolled in a prospective cohort at Xuanwu Hospital, Capital Medical University, between July 2020 and January 2024.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
favorable functional outcome. | 6 months after discharge
  mRS score ≤2 indicates favorable functional outcome.

SECONDARY OUTCOMES:
Serious steroid complications during hospitalization | from admission to discharge (up to 4 weeks after admission)
  new-onset of the following conditions:
  * lower extremity deep vein thrombosis
  * pulmonary embolism
  * gastric or duodenal ulcers
  * spontaneous fractures, osteonecrosis
  * infections or worsening of existing infections
Serious steroids complications within 6 months after discharge | 6 months after discharge
  new-onset of the following conditions:
  * Deep vein thrombosis
  * pulmonary embolism
  * gastric or duodenal ulcers
  * spontaneous fractures, osteonecrosis
  * recurrent CVT

CONTACTS AND LOCATIONS:
Overall Officials: Jiangang Duan, MD, PhD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hu S, Gu Y, Zhao T, Zhang K, Li J, Zhou C, Song H, Liu Z, Ji X, Duan J. Steroids combined with anticoagulant in acute/subacute severe cerebral venous thrombosis. Chin Med J (Engl). 2025 Aug 5;138(15):1825-1834. doi: 10.1097/CM9.0000000000003502. Epub 2025 Mar 4. PMID 40033789